CLINICAL TRIAL: NCT01889017
Title: Generic Immunosuppressive Drugs After Lung Transplantation - a Crosssectional Observational Study by Patient Questionnaire
Brief Title: Generic Immunosuppressive Drugs After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Thomas Fuehner, MD, Hannover Medical School
Other Study IDs: V 1.0 22/05/2013
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Immunosuppressive After Lung Transplantation
Keywords: generic immunosuppressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: patient questionnaire (tablet pc based)

SUMMARY:
Extent of use of generics immunosuppressive drugs in clinical practice after lung transplantation

DETAILED DESCRIPTION:
Solid organ transplant recipients are treated with immunosuppressive drugs to prevent rejection of their grafts. The most frequently important maintenance immunosuppressive drugs in Europe are calcineurin inhibitors.

For a number of these compounds drug patents have expired in recent years and generic formulations have entered the market. There is considerable debate regarding the efficacy and safety of generic drug substitution in solid organ recipients.

ELIGIBILITY:
Inclusion Criteria:

* patients after lung transplantation (single, double or combined)
* informed consent
* patient with an immunosuppressive therapy with tacrolimus or ciclosporin

Exclusion Criteria:

* immunosuppressive therapy without calcineurin inhibitors
* need for isolation (Colonization with multi. or pan resistant organisms e.g. methicillin-resistant staph. aureus[MRSA), B. cenocepacia)
* limited German language skills or other reasons which might impair patient communication or computer handling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after lung transplantation (single, double or combined) with an immunosuppressive therapy with tacrolimus or ciclosporin
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of use of generic immunosuppressive drugs | baseline

SECONDARY OUTCOMES:
Calcineurin inhibitor through levels | baseline, retrospective 6 months
  Frequency of calcineurin inhibitor through levels in target range between generic and original immunosuppressive drugs during last 6 months
Dose of calcineurin inhibitors | baseline
  Dose of calcineurin inhibitors between generic and original immunosuppressive drugs at questionnaire
Therapy adherence | baseline
  Therapy adherence between generic and original immunosuppressive drugs. Adherence will be measured by a 5 item Likert scale covering self-monitoring, generla health perception, contacts, nutrition/exercise compliance and adherence to immunosuppression.
Satisfaction with immunosuppression | baseline
  Satisfaction with immunosuppression between generic and original immunosuppressive drugs will be measured by a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Drick N, Seeliger B, Fuge J, Tudorache I, Greer M, Welte T, Haverich A, Gottlieb J. Self-reported non-adherence to immunosuppressive medication in adult lung transplant recipients-A single-center cross-sectional study. Clin Transplant. 2018 Apr;32(4):e13214. doi: 10.1111/ctr.13214. Epub 2018 Feb 23. PMID 29380445